CLINICAL TRIAL: NCT01575431
Title: PROgenitor Cells Role in Restenosis and Progression of Coronary ATherosclerosis After Percutaneous Coronary Intervention (PROCREATION) Study
Brief Title: Progenitor Cells Role in Restenosis and Atherosclerosis
Acronym: PROCREATION
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Assistant Professor, University of Roma La Sapienza
Other Study IDs: 199/2012/D
Record Dates: First submitted 2012-04-06; First posted 2012-04-11 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; endothelial progenitor cells
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stable angina: Patients who undergo an elective and successful single or multivessel percutaneous coronary intervention can be considered for the study.

SUMMARY:
The aim of this study is to prospectively investigate the relationship of circulating endothelial progenitor cells at time of percutaneous coronary intervention to the subsequent development of in-stent restenosis or progression of coronary atherosclerosis.

DETAILED DESCRIPTION:
Research on stem cells has identified a population of bone marrow-derived cells, called circulating endothelial progenitor cells (EPCs), that incorporate into sites of neovascularization and are home to sites of endothelial denudation thus contributing to the maintenance of vascular homeostasis.

Although extensive work has been conducted to verify if EPCs impairment plays a key role in coronary atherogenesis, it is still matter of debate if the extension and severity of coronary artery disease are associated with reduced or increased numbers of EPCs, as it remains unclear if these cells exert favorable or unfavorable effects at sites of percutaneous coronary intervention (PCI). One should consider, however, that most previous investigations have been hampered by discordant definitions of EPCs and by different timing of EPCs sampling, thus determining much uncertainty on the role of EPCs in restenosis and atherosclerosis progression. Furthermore, development of de novo lesions and post-PCI restenosis, which are pathophysiologically dissimilar, have not been examined concomitantly and serially over time.

Accordingly, the aim of this study is to carry out the first prospective assessment of the significance of subpopulations of circulating EPCs in the subsequent occurrence of restenosis or progression of coronary atherosclerosis after PCI. To this end, a pool of EPCs subtypes that are suggested to play some role in atherosclerosis is measured in a homogenous population of candidates to PCI. At variance with previous work, counts of EPCs are obtained in baseline conditions before PCI in order to avoid the confounding effect that the procedure exerts on EPCs.

ELIGIBILITY:
Inclusion Criteria:

* evidence of complete revascularization of clinically important stenoses by PCI
* willing to undergo 8-month control angiography.

Exclusion Criteria:

* in-hospital death after PCI
* myocardial infarction during follow-up to exclude potential subacute stent
* unstable angina
* any increase in creatine kinase-myocardial band, troponin I, myoglobin, or liver enzymes above upper normal limit before PCI
* left ventricular ejection fraction<30%
* renal failure with creatinine>2 mg/dl
* treatment with statins at referral

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patient sampling
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Results of the 1-year follow-up coronary angiography | Up to 1 year
  On the basis of the results of the 1-year follow-up coronary angiography, it will be possible to group patients in those with in-stent restenosis and those with progression of coronary atherosclerosis. Thereafter, numbers of endothelial progenitor cells at time of percutaneous coronary intervention will be compared between the two groups.

SECONDARY OUTCOMES:
Results of the 5-year clinical follow-up | Up to 5 years
  On the basis of the results of the 5-year clinical follow-up period, it will be possible to group patients in those with favorable outcome and those with a poor prognosis. Thereafter, numbers of endothelial progenitor cells at time of percutaneous coronary intervention will be compared between the two groups.
Results of the 10-year clinical follow-up | Up to 10 years
  On the basis of the results of the 10-year clinical follow-up period, it will be possible to group patients in those with favorable outcome and those with a poor prognosis. Thereafter, numbers of endothelial progenitor cells at time of percutaneous coronary intervention will be compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Pelliccia, MD, Principal Investigator — University La Sapienza
Locations (1):
- University La Sapienza, Rome, Italy

REFERENCES:
- [Derived] Pelliccia F, Pasceri V, Moretti A, Tanzilli G, Speciale G, Gaudio C. Endothelial progenitor cells predict long-term outcome in patients with coronary artery disease: Ten-year follow-up of the PROCREATION extended study. Int J Cardiol. 2020 Nov 1;318:123-125. doi: 10.1016/j.ijcard.2020.06.002. Epub 2020 Jun 6. PMID 32522679
- [Derived] Pelliccia F, Pasceri V, Rosano G, Pristipino C, Roncella A, Speciale G, Pannarale G, Schiariti M, Greco C, Gaudio C. Endothelial progenitor cells predict long-term prognosis in patients with stable angina treated with percutaneous coronary intervention: five-year follow-up of the PROCREATION study. Circ J. 2013;77(7):1728-35. doi: 10.1253/circj.cj-12-1608. Epub 2013 Apr 11. PMID 23575363